CLINICAL TRIAL: NCT05031221
Title: A Proof-of-Concept Study Examining the Addition of Yoga to a Behavioral Weight Loss Intervention on Energy Balance and Health-Related Outcomes
Brief Title: Feasibility and Impact of Yoga in Obesity
Acronym: SYNERGY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-3690
Record Dates: First submitted 2021-07-29; First posted 2021-09-01 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Yoga; Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Proof-of-Concept, single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga + behavioral weight loss (Experimental): In person and virtual yoga + 150 minutes of moderate-to-vigorous physical activity/week + weekly instruction on dietary strategies for weight loss
  Interventions: Behavioral: Yoga + behavioral weight loss

INTERVENTIONS:
Behavioral: Yoga + behavioral weight loss — A 12-week, one-arm proof-of-concept and feasibility study will be conducted at the University of Colorado Anschutz Medical Campus (CU-AMC) to assess the processes critical for the success of future randomized trials including: a) Evaluating the feasibility and acceptability of adding a multi-component yoga program to a standard BWL intervention and b) Examining pre-post changes in relevant clinical/cardiometabolic, psychological, and energy balance/behavioral outcomes to inform the design of future trials. Participants will receive a comprehensive, group-based BWL intervention consistent with current guidelines for obesity treatment and a carefully designed multi-component yoga intervention delivered through pre-recorded videos delivered through a cloud-based platform that will be completed in-person and at-home (BWL+yoga).

SUMMARY:
Yoga may confer health benefits in people with overweight or obesity that enhance weight loss and weight loss maintenance. This study aims to investigate the feasibility of integrating yoga into an established behavioral weight loss program and describe the effects on glucose control, appetite, dietary intake, physical activity, and psychological health.

DETAILED DESCRIPTION:
Innovative approaches to improve long-term behavioral weight loss (BWL) program outcomes are critically needed. Current BWL programs typically produce modest (~5-10%) short-term (~6 month) weight loss, but substantial weight regain by 1-year is common and well-documented. There has been a growing interest in examining the effects of yoga on weight loss and cardio-metabolic disease risk among adults with overweight, obesity, metabolic syndrome, pre-diabetes, and diabetes. Overall, results are somewhat promising, but reviews and meta-analyses all conclude that existing studies suffer from significant methodological shortcomings. Moreover, yoga is broadly, variably, and often incorrectly defined, reflecting how key aspects of traditional yoga practice, with specific mind, body, and breath-based practices were lost in translation when yoga was commercially adopted as a form of exercise in the West. These key aspects warrant inclusion in yoga intervention research.

The overall objectives of the proposed research are to 1) Evaluate the feasibility and acceptability of adding a 12-week traditional, multi-component yoga program to a standard BWL intervention (BWL+yoga), and 2) Explore changes in clinical/cardiometabolic, psychological, and energy balance/behavioral measures relevant for reducing cardio-metabolic disease risk. The yoga intervention was developed in collaboration with a world-renowned expert in traditional yoga practices following three decades of dedicated study, practice, and teaching (Mr. Paul Dallaghan). The program includes specific postures (asana), breathing (pranayama), and meditation (inner focus) techniques performed with an underlying focus on self-awareness delivered in-person and virtually. These specific techniques have been practiced historically and described for their benefits in the original Sanskrit teachings but are often excluded from yoga programs developed in the West. The overarching hypotheses are that these specific Hatha (body-breath) and Pantanjala (mind) yoga practices will be feasible in the context of a BWL, will support the adoption of changes in diet and physical activity, and improve mental and physical health.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-55
* Body mass index (BMI) 27-45 kg/m2
* Live or work within 30 miles of the University of Colorado Anschutz Health and Wellness Center
* Passing medical and physical screening
* Agree to fast for 12 hours before the baseline and follow-up visits
* Sedentary: defined as <150 minutes per week of voluntary exercise at moderate intensity or greater and < 60 min per day of total habitual PA (i.e. work related, transportation related) at moderate intensity or greater, over the past 3 months.
* Not currently practicing yoga regularly over past 6 months
* Among women: Not currently pregnant or lactating, not planning to become pregnant in the next 12 weeks
* English speaking, as the intervention will be delivered in English

Exclusion Criteria:

* Diastolic blood pressure > 100 mm HG or systolic blood pressure > 160 mm HG
* Resting heart rate >100
* Diabetes (fasting glucose ≥126 mg/dL or Hemoglobin A1C ≥6.5%)
* Undiagnosed hypo- or hyper-thyroidism (TSH outside of the normal range) or history of uncontrolled thyroid disorder.
* Abnormal values of: hematocrit, white blood cell count or platelets
* Triglycerides > 400 mg/dL
* LDL cholesterol >200 mg/dL
* Abnormal resting electrocardiogram (ECG)
* Presence or history of any self-reported metabolic or chronic health problems which would affect appetite, food intake, energy metabolism, or ability to optimally participate in the exercise component
* Significant self-reported pulmonary disorders including: chronic obstructive pulmonary disease (COPD), interstitial lung disease, cystic fibrosis, or uncontrolled asthma.
* Self-reported symptoms suggestive of CVD: chest pain, shortness of breath at rest or with mild exertion, syncope.
* Regular use of prescription or over-the-counter medications known to significantly impact appetite, weight, or energy metabolism
* Regular use of systemic steroids (other than Oral Contraceptive Pills).
* Regular use of obesity pharmacotherapeutic agents within the last 6 months.
* Previous obesity treatment with surgery or weight loss device
* Current alcohol or substance abuse
* Nicotine use (past 6 months)
* History of clinically diagnosed eating disorders including anorexia nervosa, bulimia, binge eating disorder.
* Current severe depression or history of severe depression within the previous year
* History of other significant psychiatric illness (e.g. psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the Study MD would interfere with ability to adhere to dietary or exercise interventions.
* Currently participating in or planning to participate in any formal weight loss or physical activity programs or clinical trials.
* Participation in a weight loss program using the Colorado Weigh curriculum within the past 3 years
* Weight loss >5kg in past 3 months for any reason except post-partum weight loss
* Weight loss of >50 lbs in past 3 years for any reason except post-partum weight loss.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Enrollment | 12 weeks before intervention initiation
  Ability to enroll 12-20 participants
Retention | At intervention completion (12 weeks)
  Attrition >20%
Collection of secondary outcome measures at baseline | Baseline (week 0)
  Percent completion of the cardiometabolic, psychological, and energy balance outcome measures
Collection of secondary outcome measures at follow-up | Intervention completion (12 weeks)
  Percent completion of the cardiometabolic, psychological, and energy balance outcome measures
Acceptability during the intervention | Week 6
  Participant satisfaction with the intervention on a 1-10 Likert scale
Acceptability after the intervention | Week 12
  Participant satisfaction with the intervention on a 1-10 Likert scale
Adherence | Weekly during the 12 week intervention
  Percent completion of intervention sessions
Adverse events (intervention safety) | Weekly during the 12-week intervention
  Study-related adverse events

SECONDARY OUTCOMES:
Body weight change | Week 0 and 12
  Body weight in kg
Resting metabolic rate (RMR) change | Week 0 and 12
  RMR in kcal/day
Body composition change | Week 0 and 12
  Fat mass and fat-free mass as measured by dual X-ray absorptiometry
Glucose tolerance change | Week 0 and 12
  2-hour oral glucose tolerance
Cardiometabolic health change | Week 0 and 12
  As measured by cholesterol, triglycerides, high- and low-density lipoproteins
Heart rate variability change | Week 0 and 12
  As measured by a 12-minute sit to stand protocol with heart rate monitor

CONTACTS AND LOCATIONS:
Overall Officials: Ann E Caldwell, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No